CLINICAL TRIAL: NCT07088536
Title: Occupational Situation of Patients With Urological Diseases and Return to Work in Patients Undergoing Major Uro-Oncological Operations and Procedures for Urinary Tract Stones
Brief Title: Occupational Situation and Return to Work of Urological Patients
Acronym: OCCURORTW
Status: Not yet recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Anna K. Czech, MD, Principal Investigator, Jagiellonian University
Other Study IDs: OCC-URO-RTW-ONCO-LITH
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Bladder Cancer; Prostate Cancer; Renal Cancer; Urinary Stones
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms; Kidney Neoplasms; Urinary Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to the Department of Urology and Oncological Urology over a 6-month period: Adult patients (≥18 years) admitted over a 6-month period to the Department of Urology and Oncological Urology, University Hospital in Kraków, Poland, including a subset of occupationally active individuals undergoing major uro-oncological surgeries or procedures for urinary tract stones.
  Interventions: Other: Occupational Status Survey and Telephone Follow-up and Quality-of-Life Assessment in a subset of patients

INTERVENTIONS:
Other: Occupational Status Survey and Telephone Follow-up and Quality-of-Life Assessment in a subset of patients — Collection of demographic, employment, and clinical data at hospital admission, with additional EQ-5D-5L quality-of-life questionnaire and telephone follow-up for occupationally active patients undergoing major uro-oncological surgeries or urinary tract stone procedures.

SUMMARY:
This study will examine the work status of all adult patients admitted over a 6-month period to the University Hospital in Kraków, Poland, for treatment of urological diseases. All admitted patients will be surveyed about their job situation. Patients who are occupationally active and undergoing major oncological surgeries (such as radical cystectomy, prostatectomy, or nephrectomy) or procedures for urinary tract stones will also complete a quality-of-life questionnaire and be followed up by phone at 3 and 6 months. The goal is to learn how treatment affects patients' ability to return to work and their well-being, to help guide support and rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years) admitted to the Department of Urology and Oncological Urology, University Hospital in Kraków, during the 6-month study period.
2. For the prospective follow-up cohort:

   1. Occupationally active (employed) at baseline.
   2. Undergoing major uro-oncological surgery (e.g., radical cystectomy, radical prostatectomy, nephrectomy) or a procedure for urinary tract stones (e.g., ureterorenoscopy, percutaneous nephrolithotripsy).
3. Able and willing to provide written informed consent.

Exclusion Criteria:

1. Patients unwilling or unable to provide informed consent.
2. Patients who are unemployed or retired at baseline (excluded from the prospective follow-up cohort but included in the baseline cross-sectional survey).
3. Patients not undergoing major uro-oncological surgery or urinary tract stone procedures (for the prospective follow-up cohort).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients admitted over a 6-month period to the Department of Urology and Oncological Urology at the University Hospital in Kraków, an academic tertiary care center in Poland. As this is a uro-oncological department, patients with urological cancers are likely to be overrepresented. The population includes individuals hospitalized for a range of urological diseases, with a subset of occupationally active patients undergoing major uro-oncological surgeries or procedures for urinary tract stones. Participants represent a typical tertiary referral population treated for both malignant and benign urological conditions.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-07-21 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Occupational Status of Patients With Urological Diseases | At hospital admission (baseline), and at 3 and 6 months for the prospective cohort
  Descriptive assessment of employment categories (employed, unemployed, on disability, retired) among all admitted patients, and changes in employment status over time for occupationally active patients undergoing major surgeries or stone-related procedures.
Return to Work Rate in Occupationally Active Patients Undergoing Major Uro-Oncological Surgeries | 3 months and 6 months after surgery
  Proportion of employed patients at baseline who resume or maintain work following radical cystectomy, radical prostatectomy, radical or partial nephrectomy, or nephroureterectomy.
Return to Work Rate in Occupationally Active Patients Undergoing Procedures for Urinary Tract Stones | 3 months and 6 months after procedure
  Proportion of employed patients at baseline who resume or maintain work following ureterorenoscopy or percutaneous nephrolithotripsy.

SECONDARY OUTCOMES:
Change in Quality of Life in Occupationally Active Patients Undergoing Major Uro-Oncological Surgeries (EQ-5D-5L Score) | Baseline, 3 months, and 6 months
Change in Quality of Life in Occupationally Active Patients Undergoing Procedures for Urinary Tract Stones (EQ-5D-5L Score) | Baseline, 3 months, and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jagiellonian University Medical College, Krakow, Malopolska, Poland

IPD SHARING:
Plan to Share IPD: Undecided